CLINICAL TRIAL: NCT04352218
Title: Novel Compliant Scaffold With Specific Design for the Treatment of Non-thrombotic Stenosis of Internal Jugular Veins in Patients With Chronic Headache Poor Responder to Best Medical Therapy
Brief Title: Safety Profile of PETALO CVS in the Treatment of Non-thrombotic Internal Jugular Vein Stenosis and Chronic Headache
Acronym: PETALO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, PIERFRANCESCO VEROUX, Professor of vascular and transplantation surgery, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CO-2018-12367503
Record Dates: First submitted 2020-02-25; First posted 2020-04-20 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Headache; Jugular Vein Occlusion
Keywords: headache; internal jugular vein obstructive disease and malformation; PTA; Stenting
MeSH Terms: conditions — Headache; Congenital Abnormalities | interventions — Angioplasty

STUDY DESIGN:
Intervention Model Description: To prospective collect and assess safety and efficacy data on the "Petalo trial" in the treatment of patients with non-thrombotic internal jugular vein stenosis and chronic headache poor responder to best medical therapy.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTA Percutaneous Transluminal Angioplasty (Active Comparator): Percutaneous Transluminal Angioplasty of internal jugular vein non-thrombotic stenosis in patients with chronic headache
  Interventions: Procedure: Percutaneous Transluminal Angioplasty (PTA)
- PTA + Stenting using "Petalo stent" (Experimental): Percutaneous Transluminal Angioplasty + Stenting of internal jugular vein non-thrombotic stenosis in patients with chronic headache
  Interventions: Device: PTA + Stenting using "Petalo stent"

INTERVENTIONS:
Device: PTA + Stenting using "Petalo stent" — PTA and Petalo's Stenting are a minimally invasive endovascular procedures, performed by a percutaneous access to the common femoral vein under local anesthesia and Duplex Ultrasound Guidance.
  Other Names: Petalo's stenting of Internal Jugular Veins
  Arms: PTA + Stenting using "Petalo stent"
Procedure: Percutaneous Transluminal Angioplasty (PTA) — PTA is a minimally invasive endovascular procedure, performed by a percutaneous access to the common femoral vein under local anesthesia and Duplex Ultrasound Guidance.
  Other Names: Venoplasty of Internal Jugular Veins
  Arms: PTA Percutaneous Transluminal Angioplasty

SUMMARY:
The purpose of the study is to assess, as first stage, the safety profile of an innovative venous- oriented device (Petalo CVS) in the treatment of patients with non-thrombotic internal jugular vein stenosis and chronic headache resistant to best medical therapy.

After Stage 1, a second stage will be conducted to evaluate the preliminary efficacy.

DETAILED DESCRIPTION:
Chronic headache is a disabling neurologic condition that affects 2-3 % of the general population. According to Headache Classification Committee of the International Headache Society, the chronic headache is defined as of at least one headache episode for 15 days a month, with at least eight days a month on which their headaches and associated symptoms meet diagnostic criteria. It is a neurologic condition characterized by attacks of headache, hypersensitivity to visual, auditory, olfactory, and cutaneous stimuli, nausea and vomiting.

Chronic migraine is common, often affects people during their most productive years of life, exerts substantial individual and societal costs, and is associated with numerous comorbid disorders. Idiopathic intracranial hypertension (IIH) has been involved in the development of chronic headache. In most of cases, IIH and chronic headache have been associated with a stenosis of the internal jugular vein (IJV). Some studies have shown that IJV compression aggravates the severity of migraine and has a possible role in the pathophysiology of migraine. Moreover, patients with migraine have less compliant IJV, which makes them susceptible to cerebral venous hypertension; these veins are more likely to develop and transmit venous hypertension caused by the increased venous blood volume during IJV compression. So, it cannot be excluded that an obstruction of the venous blood flow can lead to an increase in intracranial venous pressure and, consequently, a state of latent intracranial hypertension which justifies the chronicity of the headache. Moreover, the absence of alteration of the intracranial venous blood flow and the elevated intracranial pressure are found in about half of patients with chronic primary headache.

Based on this, among the risk factors of migraine chronicity, IIH has been evaluated like a risk factor for headache chronicity to overlap of clinical manifestations, such as persistent or high frequency headache, allodynia and to share of some factors (female sex, obesity and sleep disorders) and to the common therapeutic response to topiramate. In patients with chronic headache and IIH, a stenosis at the junction of the transverse and sigmoid sinuses has been recognized through venography but, recently, the role of isolated non-thrombotic IJV stenosis in IIH has gained a vested interest. Recent studies suggest that non-thrombotic stenosis of IJV may worsen the headache clinical severity, suggesting a possible causative role in the pathogenesis of chronic headache. It is demonstrated that the intervention of percutaneous transluminal angioplasty (PTA) was associated with a sustained improvement in clinical symptoms of patients with persistent headaches and concomitant obstructive disease of the IJV.

Balloon angioplasty and endovascular stenting of dural venous sinus stenosis in patients with IIH is a newer and actively debated treatment and has recently gained popularity. Initial studies indicate that it reduces headache in 60-88% of patients but carries 2% risk for significant morbidity and mortality.

For these reasons, given the promising risk- benefit ratio, these two therapeutics options have become an accepted treatment modality characterized by a low patency and clinical improvement rates.

Bavera et a in a prospective investigation involving 366 patients who underwent PTA and were subsequently interviewed by an independent assessor and followed up for 4 years, found improvements respectively in 98.6% of patients with headache and in 98.5% of cases with associated chronic fatigue. This latter symptom was also investigated longitudinally using two validated scales and an independent non-blinded assessor, who reported significant improvements one year after the procedure.

Furthermore, there is abundant evidence linking headaches with obstruction of the cerebral venous drainage pathways suggesting that PTA might be an effective intervention for patients suffering from persistent headaches. The endovascular treatments of non-thrombotic IJV stenosis like balloon venoplasty and stenting have been proven to provide a significant short-term improvement of IIH and related headache and a good efficacy profile with no immediate increase of risk, but data on long-term outcome are not satisfactory due to the high rate of recurrence. This suggests that PTA might be a useful intervention for treating patients with persistent headaches and concomitant obstructive disease of the IJV and that a more adequate treatment may be more appropriate rather than restenosis or recurrence. Venous stenting has emerged as an attractive therapy with the potential of addressing the intracranial pressure elevation-associated clinical issues from etiological level, particularly after medical failure. The complications of stenting such as ipsilateral headache, restenosis, intra-stent thrombosis have been demonstrated in the settings of intracranial sinus obstruction, but very few studies investigated the role and efficacy of IJV stenting in the treatment of intracranical hypertension and headache. In a recent study, the investigator found a subset of patients with presumed IIH with isolated IJV stenosis, which improved significantly their clinical symptoms (headache, tinnitus) after stenting of the IJV. The current design of stents for the venous system, however, shows improved and continuous radial force and resistance to compression. The increasing diameter of vessel toward the heart requires an oversized stent diameter to avoid migration, and this could determine the loss of the physiological compliance of the vein.

The purpose of this study is to assess the safety profile of an innovative venous-oriented device (Petalo CVS) in the treatment of patients with non-thrombotic internal jugular vein stenosis and chronic headache resistant to best medical therapy. This innovative device (Petalo CVS) has already been evaluated in an animal model in a pre-clinical study to test the safety and efficacy and has been documented a favourable safety profile of Petalo CVS.

The device Petalo CVS has been designed with full consideration of the collapsible nature of the vein, which is responsible for great variation in venous capacity with little change in venous pressure. Petalo CVS was developed considering the delicate and elastic properties of the venous wall. It has a tubular concave shape with 4 support modules joined by transverse bridges. The modules are oriented longitudinally and extend along the entire length of the device's body. The concavity of the four modules is oriented toward the vein wall. The support modules are internally empty, without bridges or other internal elements, to minimize the metal structure. Two transversal bridges join the support modules in the central part of the body, leaving the extremity of the modules free and open. The joined bridges enhance the conformability of the device and reduce the radial force. The concave shape of the support modules was studied to reduce the contact between the device and vein wall, with the aim of decreasing inflammatory. In particular, Petalo CVS was evaluated in an animal model. Twelve healthy pigs weighing 90kg were used to test it. The devices were implanted into the IJVs using a femoral vein percutaneous approach. The safety profile including the success rate of device releasing, anchoring, and positioning was evaluated immediately. Fracture, migration, primary patency, and endothelial response were assessed at 1, 2, 3, and 6 months after the study procedure. A total of 32 devices were successfully released in both IJV. No procedure -or device- related complications were reported, and all pigs successfully completed the different scheduled follow-up periods. The primary patency rate was 100%, and no fracture or migration of the device into the brachiocephalic trunk was reported. Histological examination revealed only minimal lesions with minimal or absent inflammatory reaction surrounding the incorporated metallic rods. So, this porcine model study showed a promising safety and efficacy profile of Petalo CVS.

This suggests that the particular shape and configuration of this device will assure a low rate of complications and satisfactory long-term outcomes.

Risks of venous stenting of internal jugular vein in patients with chronic headache are not well known. However, the expertise of the research group in the endovascular procedures and the shape and configuration of this device will probably determine a low rate of procedure-related complications. Long-term complications, such as thrombosis of the stent, are not well known, but the investigator's preliminary data on the animal model are encouraging.

It has been demonstrated that Petalo CVS promoted only minimal response of the vein wall, with a primary patency of 100% and the patency of the target veins was maintained without the need of any specific anticoagulant therapy.

Moreover, it is possible that not all patients with chronic headache will be suitable for venous stenting, due to unfavourable anatomy of internal jugular vein. Previous studies demonstrated that younger patients with transversal endoluminal defects are more likely to experience a significant improvement in IJV outflow after venous angioplasty, whereas in older patients with IJV hypoplasia or longitudinal endoluminal defects, angioplasty is likely to have only a limited effect. In these patients it is likely that venous stenting will have a limited efficacy and the procedure will be evaluated on a case-by-case analysis.

In general, it is expected a negligible rate of procedure-related complications such as collapse and migration to the heart.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥ 18
* Patients undergoing Echo color Doppler ultrasound with unilateral or bilateral non-thrombotic stenosis > 50% of IJV
* Patients suffering from headache not responsive to two medical treatments with diagnosis of chronic migraine or chronic tension-type headache according to the criteria of the International Classification of Headache Disorders (ICHD-3 beta).
* Subject able to comprehend the full nature and purpose of the study, including possible risks and side effects; able to co-operate with the Investigator and to comply with the requirements of the entire study.
* Subject available for the whole study period and gave written informed consent prior to inclusion in the study

Exclusion Criteria:

* Patients with unilateral or bilateral thrombosis stenosis of IJV.
* Patients with severe hypoplasia of IJV with diameter < 5mm.
* Presence of pacemaker.
* Dural venous sinus stenosis > 50%
* Documented severe intolerance to iodinated contrast medium.
* Non-compliance with pharmacological treatment
* Intracranial abnormalities such as tumor, abscess and vascular malformation.
* Severe hematological, hepatic or renal dysfunction (end-stage renal disease on dialysis will not be a contraindication).
* Life expectancy < 1 year
* Known or potential hypersensitivity to anticoagulant or antiplatelet drugs or one of the components and/or history of allergic reactions in general, which the Investigator considers important for study participation.
* Any evidence of severe or uncontrolled systemic diseases, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardies compliance with the protocol
* Females of childbearing potential will be excluded from participation in the study if they meet any one of the following conditions:
* are currently pregnant or,
* have a positive result on the urine pregnancy test or,
* intend to become pregnant during the study treatment period or, • are breast-feeding or,
* not willing to use highly effective birth control measures during the entire course of the study treatment period
* History of alcohol or drug abuse
* Enrollment in another study protocol within 30 days prior to randomization
* Any other significant disorders, which, in the opinion of the investigator, may influence the participation in the study or affect study result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Safety: Device related adverse events | 12 months
  The safety is assessed by a composite of freedom from device migration and fracture, and rupture and bleeding of the target vein within 12 months post-index procedure.
  1. Migration is defined as the displacement of the investigational device from the site of stenotic IJV tract towards the brain or anonymous trunk and right atrium and is investigated by X-radiations, DUS and CTA (if needed) through 30 days.
  2. Fracture of the Petalo's scaffold is defined as the rupture of the main modules or the bridge connections evaluated by X-radiations and CTA of the neck through 30, 90, 180 and 360 days.
  3. Bleeding is defined as a perforation of the target IJV determining an hematoma in the neck at the site of IJV stenting, and is investigated by DUS and CTA through 30, 90, 180 and 360 days.
Efficacy: Stent delivery and Primary Patency | 12 months
  1. Successful delivery and positioning of the Petalo CVS stent are defined as the precise delivery of investigational device at the site of stenotic Internal Jugular vein tract, evaluated by X-radiations, and DUS examinations through 30 days post-index procedure;
  2. Primary patency of Petalo's stent and of the target internal jugular vein is defined as freedom from stenosis > 70% of the investigational medical device and of target vein investigated by Duplex Ultrasound and CTA (in case of stenosis), through 30, 90, 180 and 360 days post-index procedure.

SECONDARY OUTCOMES:
Chronic Migraine is assessed by "Migraine Disability Assessment Score" (MIDAS). | 12 months
  The questionnaire "Migraine Disability Assessment Score" MIDAS is administered before the index procedure, and through 1, 3, 6, 12 months. The severity of migraine is defined as the following scores:
  1. Little or No Disability: 0-5 score;
  2. Mild Disability: 6-10 score;
  3. Moderate Disability:11-20 score;
  4. Severe Disability: > 20.
Major adverse events: composite of freedom from device and procedure-related mortality | 12 months
  MAEs is defined as all-cause mortality, and thrombosis at the target lesion site.
  1. All-cause mortality are assessed and documented at 30 days, 6, 12 months.
  2. Thrombosis is defined as the complete occlusion of the Petalo stent at the target lesion site, documented by DUS investigation at 30 days, 6, 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Veroux Pierfrancesco, MD, Principal Investigator — University of Catania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwedt TJ. Chronic migraine. BMJ. 2014 Mar 24;348:g1416. doi: 10.1136/bmj.g1416. PMID 24662044
- [Background] Beggs CB, Giaquinta A, Veroux M, De Marco E, Mociskyte D, Veroux P. Mid-term sustained relief from headaches after balloon angioplasty of the internal jugular veins in patients with multiple sclerosis. PLoS One. 2018 Jan 23;13(1):e0191534. doi: 10.1371/journal.pone.0191534. eCollection 2018. PMID 29360844
- [Background] Jensen RH, Radojicic A, Yri H. The diagnosis and management of idiopathic intracranial hypertension and the associated headache. Ther Adv Neurol Disord. 2016 Jul;9(4):317-26. doi: 10.1177/1756285616635987. Epub 2016 Mar 21. PMID 27366239
- [Background] Wall M. Update on Idiopathic Intracranial Hypertension. Neurol Clin. 2017 Feb;35(1):45-57. doi: 10.1016/j.ncl.2016.08.004. PMID 27886895
- [Background] Zhou D, Meng R, Zhang X, Guo L, Li S, Wu W, Duan J, Song H, Ding Y, Ji X. Intracranial hypertension induced by internal jugular vein stenosis can be resolved by stenting. Eur J Neurol. 2018 Feb;25(2):365-e13. doi: 10.1111/ene.13512. Epub 2017 Dec 7. PMID 29114973
- [Background] Bavera, M. May symptoms of chronic cerebrospinal venous insufficiency be improved by venous angioplasty? An independent 4-year follow up on 366 cases," Veins & Lymphatics, vol. 4, p. 5400, 2015
- [Background] Bono F, Messina D, Giliberto C, Cristiano D, Broussard G, D'Asero S, Condino F, Mangone L, Mastrandrea C, Fera F, Quattrone A. Bilateral transverse sinus stenosis and idiopathic intracranial hypertension without papilledema in chronic tension-type headache. J Neurol. 2008 Jun;255(6):807-12. doi: 10.1007/s00415-008-0676-2. Epub 2008 May 6. PMID 18458863
- [Background] Chung CP, Chao AC, Hsu HY, Lin SJ, Hu HH. Decreased jugular venous distensibility in migraine. Ultrasound Med Biol. 2010 Jan;36(1):11-6. doi: 10.1016/j.ultrasmedbio.2009.08.007. PMID 19900748
- [Background] Zamboni P, Galeotti R, Menegatti E, Malagoni AM, Gianesini S, Bartolomei I, Mascoli F, Salvi F. A prospective open-label study of endovascular treatment of chronic cerebrospinal venous insufficiency. J Vasc Surg. 2009 Dec;50(6):1348-58.e1-3. doi: 10.1016/j.jvs.2009.07.096. PMID 19958985
- [Background] Zamboni P, Galeotti R, Weinstock-Guttman B, Kennedy C, Salvi F, Zivadinov R. Venous angioplasty in patients with multiple sclerosis: results of a pilot study. Eur J Vasc Endovasc Surg. 2012 Jan;43(1):116-22. doi: 10.1016/j.ejvs.2011.03.035. Epub 2011 Aug 11. PMID 21839654
- [Background] Lee BB, Baumgartner I, Berlien P, Bianchini G, Burrows P, Gloviczki P, Huang Y, Laredo J, Loose DA, Markovic J, Mattassi R, Parsi K, Rabe E, Rosenblatt M, Shortell C, Stillo F, Vaghi M, Villavicencio L, Zamboni P. Guideline. Diagnosis and treatment of venous malformations. consensus document of the international union of phlebology (iup): updated-2013. Int Angiol. 2014 Jun 10. Online ahead of print. PMID 24961611
- [Background] Veroux P, Giaquinta A, Virgilio C, Zani DD, Ravasio G, Ardita V, Secchiero P, Scanziani E, Zamboni P, Veroux M. Novel Compliant Scaffold with Specific Design for Venous System: Results of a Porcine Model Study. Biomed Res Int. 2018 Jan 31;2018:7312315. doi: 10.1155/2018/7312315. eCollection 2018. PMID 29662897
- [Background] Stewart WF, Lipton RB, Dowson AJ, Sawyer J. Development and testing of the Migraine Disability Assessment (MIDAS) Questionnaire to assess headache-related disability. Neurology. 2001;56(6 Suppl 1):S20-8. doi: 10.1212/wnl.56.suppl_1.s20. PMID 11294956
- [Background] Zamboni P, Giaquinta A, Rimondi E, Pedriali M, Scanziani E, Riccaboni P, Veroux M, Secchiero P, Veroux P. A novel endovenous scaffold for the treatment of chronic venous obstruction in a porcine model: Histological and ultrastructural assessment. Phlebology. 2019 Jun;34(5):336-346. doi: 10.1177/0268355518805686. Epub 2018 Oct 18. PMID 30336762